CLINICAL TRIAL: NCT00291226
Title: Glycine vs Placebo for the Schizophrenia Prodrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Glytech, Inc (Industry); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0502027440
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2016-11

CONDITIONS: Schizophrenia Prodrome
Keywords: schizophrenia prodrome
MeSH Terms: interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycine (Experimental): Glycine dosing was fixed at an initial dose of 0.2 g/kg q.h.s for 3 days, then 0.2 g/kg b.i.d. for 4 days, then 0.2 g/kg in the a.m. and 0.4 g/kg in the p.m. for 4 days, and finally 0.4 g/kg b.i.d. Subjects weighing > 100 kg were limited to a total daily dose of 80 g daily. Glycine was dispensed under IND 33,515 (DCJ).
  Interventions: Drug: Glycine
- Placebo Group (Placebo Comparator): Placebo was dispensed as a proprietary formulations developed by Glytech, Inc, consisting of microencapsulated sucrose. Recommended administration of the sprinkles was to spoon them onto pudding or applesauce and swallow them with minimal chewing. Since earlier product testing by Glytech revealed that a few individuals did not like the somewhat granular texture of the sprinkles, subjects could switch to a second Glytech placebo formulation, consisting of proprietary pre-flavored sugar powders to be dissolved in 8 ounces of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glycine — Glycine 0.4 g/kg bid
  Arms: Glycine
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Glycine is a natural amino acid neurotransmitter that acts as a co-agonist at NMDA receptors in brain. We hypothesize that symptoms of the schizophrenia prodrome will improve with glycine to a greater degree than with placebo.

DETAILED DESCRIPTION:
A pilot clinical trial comparing glycine to placebo in patients with the schizophrenia prodrome.

ELIGIBILITY:
Inclusion Criteria:

* meet SIPS criteria for schizophrenia prodrome

Exclusion Criteria:

* history of psychosis

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University
Locations (1):
- PRIME Clinic, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woods SW, Walsh BC, Hawkins KA, Miller TJ, Saksa JR, D'Souza DC, Pearlson GD, Javitt DC, McGlashan TH, Krystal JH. Glycine treatment of the risk syndrome for psychosis: report of two pilot studies. Eur Neuropsychopharmacol. 2013 Aug;23(8):931-40. doi: 10.1016/j.euroneuro.2012.09.008. Epub 2012 Oct 22. PMID 23089076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between March 2006 and May 2008. Potential subjects or their families or providers were informed about the symptoms of the risk syndrome for psychosis through a variety of ongoing community education efforts and were invited to call our research clinic if concerned.
Pre-assignment Details: Exclusions: 1) past or current DSM IV criteria for any lifetime psychotic disorder, 2) alcohol or drug abuse or dependence in the past three months, 3) use of antipsychotic medication in the previous three months, 4) change in dosage of any antidepressant, anxiolytic, psychostimulant, or mood stabilizer medication within eight weeks.
Groups:
- Glycine: Glycine dosing group.
- Placebo Group: Glycine and placebo dosing group.
Period: Overall Study
Arm/Group | Glycine | Placebo Group
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Glycine: Glycine dosing was fixed at an initial dose of 0.2 g/kg q.h.s for 3 days, then 0.2 g/kg b.i.d. for 4 days, then 0.2 g/kg in the a.m. and 0.4 g/kg in the p.m. for 4 days, and finally 0.4 g/kg b.i.d. Subjects weighing > 100 kg were limited to a total daily dose of 80 g daily.
  Glycine and placebo were dispensed under IND 33,515 (DCJ) as one of two proprietary formulations developed by Glytech, Inc. Dosing was initiated with small microencapsulated beads or "sprinkles" (80% glycine by weight), with placebo consisting of microencapsulated sucrose. Recommended administration of the sprinkles was to spoon them onto pudding or applesauce and swallow them with minimal chewing.
  Glycine: Glycine 0.4 g/kg bid
- Placebo Group: Glycine and placebo were dispensed under IND 33,515 (DCJ) as one of two proprietary formulations developed by Glytech, Inc. Dosing was initiated with small microencapsulated beads or "sprinkles" (80% glycine by weight), with placebo consisting of microencapsulated sucrose. Recommended administration of the sprinkles was to spoon them onto pudding or applesauce and swallow them with minimal chewing. Since earlier product testing by Glytech revealed that a few individuals did not like the somewhat granular texture of the sprinkles, subjects could switch to a second Glytech formulation, consisting of proprietary pre-flavored glycine or sugar powders to be dissolved in 8 ounces of water.
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Glycine | Placebo Group | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (0.5) | 16.5 (2.4) | 15.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Scale of Prodromal Symptoms Total Score
Description: Scale Of Prodromal Symptoms (SOPS) is a 19-item instrument. The SOPS is comprised of symptoms that are classified as falling into four pathology domains: positive, negative, disorganized and general. The scales identify and measure five attenuated positive psychotic symptoms, six negative symptoms, four disorganization symptoms and four general symptoms. These seven-point scales cover severity variance in the subpsychotic or attenuated range. Each item is scaled 0-6, with 0-2 being the normal range, 3-5 being the risk syndrome range, and 6 being severe and psychotic for the positive symptoms and very severe for the other symptoms. The higher the score, the more symptoms an individual has and is therefore negative in its interpretation. The severity of the prodromal state is judged according to the sum of the ratings from each of the SOPS items and can range from 0 to 114. Actual SOPS total scores in this study ranged from 23 to 59 across subjects at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glycine | Placebo Group
Number analyzed (Participants) | 4 | 4
units on a scale | 37.8 (15.3) | 37.5 (10.0)

2. Primary Outcome: Change in Scale of Prodromal Symptoms Total Score
Description: as for outcome 1
Time Frame: Change from Baseline at 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glycine | Placebo Group
Number analyzed (Participants) | 4 | 4
units on a scale | -5.8 (8.1) | 4.5 (9.7)

ADVERSE EVENTS:
Arm/Group | Glycine | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycine (N=4) | Placebo Group (N=4)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Sedation (Psychiatric disorders) | 0 (0) | 2 (2)
Orgasm Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Disturbed Sleep (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Mentation Impaired (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Stomach Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes